CLINICAL TRIAL: NCT01305499
Title: A Randomized Phase II Trial to Simultaneously Evaluate Two Schedules of the Histone Deacetylase Inhibitor Entinostat in Combination With 5-Azacytidine (5AC, NSC 102816) in Elderly Patients With Acute Myeloid Leukemia (AML)
Brief Title: A Trial to Evaluate Two Schedules of MS275 in Combination With 5AC in Elderly Patients With Acute Myeloid Leukemia (AML)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hetty Carraway (Other)
Responsible Party: Sponsor-Investigator, Hetty Carraway, MD, MBA, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE2914; 15-851 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A: 5AC days 1-10 / entinostat days 3, 10 (Experimental): Arm A will be given an overlapping schedule of drugs with 5AC given at 50mg/m2 subcutaneously daily for 10 days on days 1 - 10 of a 28 day cycle and entinostat given at a flat dose of 8 mg orally on days 3 and 10.
  Interventions: Drug: Entinostat days 3, 10; Drug: 5AC
- B: 5AC days 1-10 / entinostat days 10,17 (Experimental): In Arm B the agents will be administered sequentially with 5AC given at 50mg/m2 subcutaneously daily for 10 days on days 1 - 10 of a 28 day cycle followed by entinostat at a 8 mg flat dose on days 10 and 17.
  Interventions: Drug: 5AC; Drug: Entinostat days 10,17

INTERVENTIONS:
Drug: Entinostat days 3, 10 — Given orally on days 3, 10
  Other Names: MS275
  Arms: A: 5AC days 1-10 / entinostat days 3, 10
Drug: 5AC
  Other Names: 5-azacitidine
Drug: Entinostat days 10,17 — Given orally on days 10, 17
  Other Names: MS275
  Arms: B: 5AC days 1-10 / entinostat days 10,17

SUMMARY:
This research is being done to help us learn how to best use new drugs which may be active against acute myeloid leukemia (AML). Two study drugs will be tested: 5AC (5-azacitidine) and entinostat. 5AC improves blood counts in 50 - 60% of patients with MDS and has also shown promise in AML. Entinostat has undergone early testing in patients with MDS and AML. It has decreased the blast count in some patients' blood and bone marrow and has improved the blood counts in some patients. The combinations of these two classes of drugs are well tolerated and appear to work well together in laboratory tests.

A recent study at Johns Hopkins University administered 5AC and entinostat in an overlapping schedule to patients with myelodysplastic syndrome (MDS), Chronic myelomonocytic leukemia (CMMoL), and AML. The impressive results from this study have led to another phase II trial to further examine this drug combination versus 5AC alone in these patients. In this study, we want to see how the timing of when 5AC and entinostat are given affects the magnitude of the disease response.

DETAILED DESCRIPTION:
1. To estimate the major response rate (complete and partial responses by the International Working Group (IWG) response criteria) in patients with AML who are >= 60 years old and unable to tolerate or decline cytotoxic chemotherapy or patients who have relapsed despite one prior regimen and are treated with (a) 5AC 50mg/m2 subcutaneously/intravenously for 10 days on days 1 - 10 of a 28 day cycle given in combination with entinostat 8 mg (flat dose) administered orally on days 3 and10 of each cycle or (b) the same regimen of 5AC with entinostat given on days 10 and 17.
2. To estimate the overall response rate (complete, partial, and hematologic improvement- major by IWG criteria) following treatment with two different dose schedules of 5-Azacytidine and entinostat in patients with AML >= 60 years old who are unable to tolerate or decline cytotoxic chemotherapy or those who have relapsed despite one prior regimen.

The secondary objectives of the study are:

1. To identify changes in gene promoter methylation and gene expression in response to combination therapy with 5AC and entinostat and compare the dynamics and kinetics of these alterations in promoter methylation and gene re-expression in the two different dosing schedules.
2. To evaluate the effect of entinostat on the induction of hyperacetylation of histones from peripheral blood and/or bone marrow samples.
3. To evaluate changes in DNA damage in response to combination therapy using gammaH2AX determination by western blotting.
4. To evaluate immune parameters after exposure to 5AC and entinostat when given at either dosing schedule and to evaluate these in relation to clinical outcomes.
5. To evaluate duration of response.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following:

   Untreated AML in (de novo or treatment related) patients in the following categories:
   * Medical conditions that compromise the ability to give cytotoxic chemotherapy as the primary modality.
   * Patients who decline cytotoxic chemotherapy.

   Patients with AML who have relapsed despite one prior regimen
2. ECOG performance status 0, 1, or 2
3. Patients must not have untreated active infections at the time of study entry.
4. Normal organ function as defined below:

   * Creatinine < 2 mg/dl.
   * Total serum bilirubin within institutional limits unless due to hemolysis, Gilbert's syndrome, or ineffective erythropoiesis.
   * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal.
5. Life expectancy of at least three months.
6. Patients must be informed of the investigational nature of the treatment, results that might be expected, and potential toxicities. They must be able to understand and give informed written consent according to federal and institutional guidelines.
7. Declined or ineligible for potentially curative options such as allogeneic stem cell transplant.
8. No chemotherapy or study drugs for >3 weeks prior to starting study.
9. Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment. All men and women of childbearing potential must use acceptable methods of birth control throughout the study as described below:

   * Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation.
   * Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study or to abstain.

Exclusion Criteria

1. Any of the Following:

   * Treatment for acute myeloid leukemia (AML), including hematopoietic growth factors, < 3 weeks prior to study registration. Exception: Hydroxyurea may be administered to patients with WBC > 30,000/µL
   * Diagnosis of acute promyelocytic leukemia (APL)
   * Radiotherapy < 4 weeks prior to study registration
   * Failure to recover (to < grade 1) from all adverse events associated with prior therapy.
   * Valproic acid < 2 weeks prior to study registration.
   * Hypersensitivity to azacytidine, deoxyazacytidine, mannitol, entinostat or components of the entinostat tablet
   * Any advanced malignant hepatic tumor(s)
2. Prior therapy with demethylating agents for leukemia treatment within the last four months.
3. Clinical evidence of CNS or pulmonary leukostasis, disseminated intravascular coagulation, or central nervous system leukemia.
4. Serious or uncontrolled medical conditions.
5. Concurrent use of any other investigational agents.
6. Known HIV-positive patients.
7. Pregnancy or breast feeding
8. Male and female patients who are fertile who do not agree to use an effective barrier methods of birth control (i.e. abstinence) to avoid pregnancy during the study and for a minimum of 30 days after study treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To estimate the major response rate in patients with AML who are ≥ 60 years old and unable to tolerate or decline cytotoxic chemotherapy or patients who have relapsed despite one prior regimen. | Up to 15 cycles (420 days)
To estimate the overall response rate following treatment in patients with AML ≥ 60 years old who are unable to tolerate or decline cytotoxic chemotherapy or those who have relapsed despite one prior regimen. | Up to 15 cycles (420 days)

SECONDARY OUTCOMES:
To identify changes in gene promoter methylation and gene expression in response to combination therapy and compare the dynamics and kinetics of these alterations in promoter methylation and gene re-expression in the two different dosing schedules. | Up to 15 cycles (420 days)
To evaluate the effect of entinostat on the induction of hyperacetylation of histones from peripheral blood and/or bone marrow samples. | Up to 15 cycles (420 days)
To evaluate changes in DNA damage in response to combination therapy using gammaH2AX determination by western blotting. | Up to 15 cycles (420 days)
To evaluate the pharmacodynamics of 5AC and entinostat when given at either dosing schedule and to evaluate these in relation to pharmacokinetic and clinical outcomes. | Up to 15 cycles (420 days)
To evaluate duration of response. | Up to 15 cycles (420 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hetty Carraway, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Yale School of Medicine, New Haven, Connecticut
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio